CLINICAL TRIAL: NCT00372268
Title: Evaluation of the Effects of Conditioning of Insufflated Gas on the Core Temperature and the Post-operative Pain During Laparoscopic Surgery
Brief Title: Effects of Insufflated Gas on Core Temperature and Post-operative Pain During Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3621
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Laparoscopy; Pain, Postoperative; Hypothermia
Keywords: Comparison of four conditionings of the insufflated gas during laparoscopy and their consequences on the core temperature and the post-operative pain.; Women with womb pathology needing laparoscopic surgery; No emergency; Aged over 18 years
MeSH Terms: conditions — Pain, Postoperative; Hypothermia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- B (Active Comparator): Administration of ropivacaïne 0,2% by direct intra-abdominal administration at the end of the surgery
  Interventions: Device: Aeroneb® Pro (Nektar® Company)
- C (Active Comparator): Administration of ropivacaïne 0,75% by nebulization in the insufflated gas during all the surgical procedure with direct intra-abdominal administration of Nacl 0,9%
  Interventions: Device: Aeroneb® Pro (Nektar® Company)
- A (Placebo Comparator): Administration of Nacl 0,9% by nebulization in the insufflated gas during all the surgical procedure with direct intra-abdominal administration of Nacl 0,9%
  Interventions: Device: Aeroneb® Pro (Nektar® Company)
- D (Placebo Comparator): Administration of Nacl 0,9% by direct intra-abdominal administration at the end of the surgery
  Interventions: Device: Aeroneb® Pro (Nektar® Company)

INTERVENTIONS:
Device: Aeroneb® Pro (Nektar® Company) — The Aeroneb® Pro (Nektar® Company) permits cold and wet nebulization of either saline solution or ropivacaïne 0.75% (Naropeine) during the surgical procedure.
  Arms: A; C
Device: Aeroneb® Pro (Nektar® Company) — The Aeroneb® Pro (Nektar® Company) permits cold and dry nebulization without saline solution neither ropivacaïne (Naropéine) during the surgical procedure.
  Arms: B; D

SUMMARY:
During laparoscopy, administration of cold and dry carbon dioxide (CO2) leads to hypothermia. Different types of gas conditioning have been studied in order to prevent this specific hypothermia. Intra-abdominal administration of local anesthetics has also been studied in order to prevent post-operative pain. In both cases, some results have been described.

The investigators propose to evaluate in a prospective, randomized, double blind trial, the impact of 4 different types of conditioning of insufflated gas during laparoscopy for womb surgery on hypothermia prevention and post-operative pain. These 4 types of gas conditioning are:

* CO2 wet and cold with nebulized Nacl and direct intra-abdominal administration of Nacl
* CO2 wet and cold with nebulized ropivacaïne 0.75% and direct intra-abdominal administration of Nacl
* CO2 dry and cold with direct intra-abdominal administration of ropivacaïne 0.2%
* CO2 dry and cold with direct intra-abdominal administration of Nacl

The investigators use a new device (Aeroneb® Pro [Aerogen® Company]) which can wet (by nebulization) the insufflated gas and therefore permits intraperitoneal medicament administration (local anesthetics).

ELIGIBILITY:
Inclusion Criteria:

* Womb surgery by laparoscopy
* Female
* Aged over 18 years
* No emergency

Exclusion Criteria:

* Laparotomy
* Protocol rejected by the patient
* Request of the surgeon or the anesthesiologist to know the administration solution or the insufflated gas

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2006-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evolution of core temperature | From the beginning of the anesthetic procedure to the discharge of the recovery room.
Post-operative pain | From the arrival in the recovery room to the 6th post-operative day.

SECONDARY OUTCOMES:
Inflammation parameters | From the beginning of the anesthetic procedure to the end of the surgical procedure (one blood sample is done before the surgery, the second is done just after the arrival in the recovery room)
Quality of life | From the discharge of the recovery room to the 6th post-operative day
Surgical comfort | During the duration of the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DIEMUNSCH, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (3):
- France (2):
  - Sihcus-Cmco, Schiltigheim
  - Hôpital de Hautepierre, Strasbourg
- Department of Perioperative Medicine and Intensive Care - SAN GERARDO HOSPITAL, Monza, Italy

REFERENCES:
- [Result] Greib N, Schlotterbeck H, Dow WA, Joshi GP, Geny B, Diemunsch PA. An evaluation of gas humidifying devices as a means of intraperitoneal local anesthetic administration for laparoscopic surgery. Anesth Analg. 2008 Aug;107(2):549-51. doi: 10.1213/ane.0b013e318176fa1c. PMID 18633034